CLINICAL TRIAL: NCT06422780
Title: Comparison of Maternal Role Preparation and Awareness-Centred Occupational Therapy Trainings in Pregnant Women: Randomised Controlled Trial With Postpartum Follow-up
Brief Title: Comparison of Maternal Role Preparation and Awareness-Centred Occupational Therapy Trainings in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Aysenur KARAKUS, Lecturer, Çankırı Karatekin University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HÜ-ERG-AK-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Postpartum Complication
Keywords: pregnancy; postpartum period; occupational therapy; quality of life

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Maternal Role Preparation Training Group (Active Comparator): Pregnant women in the second trimester (14-27th week) will be included in the trainings.
  Interventions: Other: Maternal Role Preparation Training
- Awareness Centred Occupational Therapy Group (Active Comparator): Pregnant women in the second trimester (14-27th week) will be included in the trainings.
  Interventions: Other: Awareness Centred Occupational Therapy Group
- Control Group (No Intervention): Pregnant women in the second trimester (14-27th week) will be included in the trainings.

INTERVENTIONS:
Other: Maternal Role Preparation Training — Maternal Role Preparation Training: Maternal Role Preparation Training (MRHE) is an occupational training programme aimed at increasing the competence of first-time mothers regarding motherhood. In this four-session programme, pregnant women will be provided with written materials, face-to-face talks and practical training covering topics related to their babies (maternal attachment, training on the sensory and developmental abilities of babies) and themselves (training on adopting a new role as a mother).The sessions will be applied 2 days a week, each session 1 hour, a total of 8 weeks-16 sessions.
  Arms: Maternal Role Preparation Training Group
Other: Awareness Centred Occupational Therapy Group — Awareness Centred Occupational Therapy (FME); In FME, areas that affect the occupational performance of pregnant women in their daily lives will be identified and appropriate occupational therapy interventions will be applied. Awareness training on the applications will be given before starting the sessions. The sessions will be applied 2 days a week, each session 1 hour, a total of 8 weeks-16 sessions. Awareness training will be given before starting the sessions.
  Arms: Awareness Centred Occupational Therapy Group

SUMMARY:
The aim of this study was to compare maternal role preparation and mindfulness-centred occupational therapy trainings in pregnant women: a randomised controlled trial with postpartum follow-up.

DETAILED DESCRIPTION:
Pregnancy and postpartum are a major change and crisis process for women. Women undergo hormonal, vascular, anatomical, physiological, and psychological changes for 40 weeks to meet the biochemical needs of the developing fetus, maintain homeostasis, and prepare for childbirth and lactation. These changes occurring during pregnancy are necessary to protect the health of mother and baby, as well as to prepare women for childbirth and maternity.

Psychological changes that vary from trimester to trimester, accompanied by physiological changes in pregnancy. Especially in the second and third trimester, changes in the biopsychosocial balance, affecting family and work roles, taking on new responsibilities, trying to adapt to new roles and meeting the baby increased perceived depression, anxiety and stress. These physiological and psychological symptoms during pregnancy have been to adversely affect the quality of life of pregnant women. In literature, participation in meaningful and purposeful activities, which is an important indicator of quality of life, is also believed to have an impact on occupational performance during pregnancy. During pregnancy, post-partum and postpartum, the mother is expected to adapt to the physiological and psychological changes she experiences, to be able to take care of herself and her baby, to play the role of mother and to accept her baby. Physical activity levels, sleep and quality of life during pregnancy are also likely to be affected by maternal role adaptation and participation in social life. In this context, it should be taken into account that the period of pregnancy is an important milestone for the end of childbirth and the postpartum period.

Postpartum physical problems occur in 70% of women, while 17% of women are accompanied by emotional problems.Especially in the postpartum period, emotional changes have been to occur in between 24% and 89% of women with post-partum depression (PPD), between 40% and 50% of mothers and between 9% and 30% of female with anxiety. Emotional problems can also arise as a result of a mother's physical problems, such as providing baby care, creating a safe environment for the baby, communicating with the child, learning new roles, developing family sensitivity, and dealing with problems related to the baby. Therefore, the postpartum period can become a crisis life for the family, just like pregnancy.Physical and emotional symptoms may adversely affect family, work, and social life, thereby reducing quality of life. (14,15,24). Physical and emotional symptoms have also been to negatively affect the maternal bond between the mother and the baby, the mother's sense of self, occupational balance, and occupational performance.

Occupational Theraphy is a health care profession that supports an individual's ability to sustain occupational performance through various interventions and person-centric practices, helping the individual to adapt to changes that are constantly encountered within and around him. In this context, one of the interventions used to enhance pregnancy coherence is maternal role preparation training. Maternal role preparation is an occupational training that focuses on improving motherhood competence and living a successful role-to-mother harmony when the mother becomes a mother for the first time.

One of the other interventions used in occupational therapy is a person-centric occupation therapy. In today's occupational therapy interventions, person-centric practices have always been a key element. With a person-centric approach, consultants and therapists work together to identify the nature of their occupational performance problems, the focus and need of the intervention, and the consequences of the preferred treatment.

In this context, the study was planned to study tangible behavioral changes resulting from interventions in healthy pregnant women and their impact on participation in daily life activities. Our study aims to study the effectiveness of maternal role preparation training and awareness-based occupational therapy and post-partum follow-up.

This study is important for the continuation of valuable activities and roles within pregnant women's daily routines, for the development of new strategies to make them feel better during pregnancy, and for a clinically integrated approach.

ELIGIBILITY:
Inclusion criteria for pregnant women:

* 18 to 35 years of age
* Having conceived naturally
* Being between 14-27 weeks of gestation
* To be literate
* Being primiparous
* Reading and understanding Turkish
* Volunteering to participate in the study
* To have attended 80% of the trainings given

Inclusion criteria for women in the postpartum period:

* Giving birth at term
* Having a healthy newborn (newborn born at 38-42 weeks of gestation, without low birth weight, without any disease)
* Providing active care to the newborn baby with or without assistance

Exclusion criteria for pregnant women

* Having a risky pregnancy (gestational diabetes, eclampsia, pre-eclampsia, threatened preterm birth, premature rupture of membranes, placental anomalies etc.)
* Having a maternal physical anomaly
* Communication difficulties and mental deficiency
* Having a medical history of mental illness
* Having a foetal abnormality during pregnancy
* Having a disease/complication that developed during pregnancy

Exclusion criteria for women in the postpartum period:

* Experiencing a traumatic event within 6-8 weeks postpartum (loss/death of a close person, natural disasters, accident, assault)
* Stillbirth or having a baby with anomalies
* Having a baby that requires an intensive care environment in a hospital
* Mothers diagnosed with psychiatric illness (schizophrenia, depression, anxiety, panic attacks)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Nothingham Health Profile(NHP) | 3 weeks
  The Nottingham Health Profile will be used to assess the awareness of pregnant women about their own health status. The Nottingham Health Profile assesses self-perceived health status and includes subsections on pain, emotional reactions, sleep, social isolation, physical activity and energy. These sub-sections make up the more intensively used section 1, while work life, household chores, social life, home life, sexual life, interests and holidays make up section 2. Each section is scored on a scale of 0-100. In the sections consisting of questions answered yes and no, the highest score can be 0 and the lowest score can be 100 (40,41). Turkish adaptation was performed by Küçükdeveci et al. in 1997.

SECONDARY OUTCOMES:
Demographic Data Form | 1 weeks
  Physical, demographic and obstetric information of pregnant women will be recorded. In the physical information section, the height (m), body weight (kg) before pregnancy and at the time of assessment will be recorded. In the demographic information section, the age, marital status ("married" and "single"), educational status of the pregnant woman and the father, employment status ("working" and "not working") and occupation of the pregnant woman and the father will be questioned. Educational status will be recorded categorically as "only literate", "primary school", "secondary school", "high school", "associate degree", "bachelor's degree", "master's degree" and "doctorate"
Occupational Balance Questionnaire(OBQ11-T) | 3 weeks
  The validity and reliability study of the Turkish version, developed by Wagman and Hakansson (2012), was carried out by Günal et al. (2019). The test-re-test reliability ratio for the Turkish version of the scale was 0.922, with the Cronbach alpha value being 0.785. The room is a self-reporting scale that evaluates a person's occupational balance in different dimensions. It is used to measure the satisfaction a person receives from the number and variety of daily activities and to determine the occupational balance based on the results obtained. The scale consists of 11 items rated at a 4-point range ranging from 0 (I totally disagree) to 3 (I absolutely agree). The scale's total score is the sum of the individual scores given to the questions and ranges from 0-33. High scores indicate a better occupational balance.
Time Management Questionnaire(TMQ) | 3 weeks
  Time management of individuals will be evaluated by Time Management Questionnaire (TMQ) consisting of 27-items. Developed by Britton and Tesser (1991), Alay and Koçak (2002) conducted a Turkish reliability and validity study. The reliability coefficient calculated by Cronbach's alpha correlations was found to be 0.88 for Time Planning, 0.66 for Time Attitudes subscale and 0.87 for the whole scale. The ATI is an inventory with 3 subscales: 16-item Time Planning, 7-item Time Attitudes and 4-item Time Spenders. Each item is scored out of 5 and a five-point scale consisting of "always, often, sometimes, rarely and never" options is formed. In scoring, 5 is given to the answer at the end of the scale, while 1 is given to the answer on the other side of the scale. The maximum score that can be obtained from the RIQ is 135 and the minimum score is 27.
The Hospital Anxiety and Depression Scale(HADS) | 3 weeks
  Hospital Anxiety and Depression Scale (HADS): HAD was developed by Zigmond and Snaith (47) in 1983. Turkish validity and reliability of the scale was performed by Aydemir in 1997. The scale consists of 14 items. Odd numbered items in the scale investigate anxiety and even numbered items investigate depression. Seven items measure anxiety and seven items measure depression. In the Turkish validity and reliability study of the scale, the cronbach alpha coefficient was found to be 0.85 for the anxiety subscale and 0.77 for the depression subscale. In this study, the cronbach alpha values of the scale sub-dimensions were found to be 0.88 for the anxiety sub-dimension and 0.79 for the depression sub-dimension.
The Cognitive Emotion Regulation Questionnaire | 3 weeks
  It was developed by Garnefski, Kraaij, and Spinhoven (2001) and adapted into Turkish by Tuna and Bozo (2012) (50, 51). When the scale was analysed in terms of reliability, Cronbach's alpha coefficients of the subscales ranged between .68 and .86 in various populations. The five-point Likert-type scale (1= almost never, 2= rarely, 3= sometimes, 4= often, 5= almost always) consists of a total of 36 items. Each subscale consists of four items representing different emotion regulation strategies: self-blame, acceptance, rumination, perspective taking, positive refocusing, planning refocusing, positive reappraisal, catastrophising and blaming others. Subscale scores are obtained by summing the item scores corresponding to the relevant subscale and each subscale receives a score between 4 and 20. Higher scores on the subscales indicate a higher frequency of using the relevant emotion regulation strategy.
Coping Style Scales | 3 weeks
  It is a 4-point Likert-type scale that evaluates individuals' coping styles with stress (44, 45). This scale was developed by Folkman and Lazarus (1988) and Turkish reliability and validity study was conducted by Şahin and Durak (1995). Cronbach alpha internal consistency coefficients were reported to be between 0.49-0.68 for optimistic approach, 0.62-0.80 for self-confident approach, 0.64-0.73 for helpless approach, 0.47-0.72 for submissive approach and 0.45-0.47 for social support seeking factor. SBSAS consists of 5 factors: self-confident approach, helpless approach, submissive approach, optimistic approach and seeking social support. The scale is a 5-point Likert-type self-report scale consisting of 31 items. The scale includes a metric measurement from "I Never Use" (0) to "I Always Use" (4). The scores obtained from the scale vary between 0-124.
Visual Pain Scale(VPS) | 3 weeks
  The pain intensity of the pregnant women was questioned with a 10 cm visual analogue scale (VAS). In this scale, the beginning of the line indicates "no pain" (score 0) and the end of the line indicates "unbearable pain" (score 10). Pregnant women will be asked to mark the intensity of the pain they feel on the VAS. The marked point will be measured with a ruler and the results will be recorded in cm.
Visual Sleep Scale(VSS) | 3 weeks
  The degree of sleep problems of the pregnant women will be evaluated using a VAS consisting of a 10 cm line. On this 10 cm line, the pregnant women will be told that the point "0" means that there is no problem with sleep and the point "10" means a very severe sleep problem and they will be asked to mark their sleep problems on this line. The marking point will be measured with the help of a ruler and the value obtained will be recorded in cm. In addition, the total amount of sleep of the pregnant women and how much sleep they wake up at night will be questioned in hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University Occupational Therapy Department, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No